CLINICAL TRIAL: NCT03259880
Title: Searching the Best Best Prognostic Factor in Out Come Evaluation in Patients With Acute Pancreatitis Admitted at Assiut University Hospitals
Brief Title: Searching the Best Prognostic Factor in Out Come Evaluation in Patients With Acute Pancreatitis Admitted at Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fady Refaat Edwar Nasrallah (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Fady Refaat Edwar Nasrallah, internal medicine resident,Assiut University hospital, Assiut University
Organization: Assiut University (Other)
Other Study IDs: assiut university 7001
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Acute Pancreatitis
Keywords: evaluation
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute pancreatitis (AP) is rapid-onset inflammation of the pancreas that varies in severity from a self-limiting mild illness to rapidly progressive multiple organ failure. Statistics suggest that 10-20% of patients with AP develop severe AP (SAP),1 which usually has an unfavourable disease progression and is associated with a poor prognosis.

The two most common and important causes of acute pancreatitis are gallstones (40-70%) and alcohol (25-35%) Gallstone pancreatitis is usually due to an obstructing stone in the pancreatic duct near the sphincter of Oddi . In alcohol-related pancreatitis, it is believed that the acinar cells of the pancreas are susceptible to damage by ethanol and underlie the etiology of the disease . Another common cause, iatrogenic pancreatitis, may occur after endoscopic retrograde cholangiopancreatography (ERCP) in up to 5% of patients. Other etiologies of acute pancreatitis include medications, infections, trauma, hereditary, hypertriglyceridemia and autoimmune disease.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is rapid-onset inflammation of the pancreas that varies in severity from a self-limiting mild illness to rapidly progressive multiple organ failure. Statistics suggest that 10-20% of patients with AP develop severe AP (SAP),1 which usually has an unfavourable disease progression and is associated with a poor prognosis. (Banks PA, Bollen,et al.).

The two most common and important causes of acute pancreatitis are gallstones (40-70%) and alcohol (25-35%) (Tenner S et al., 2014) Gallstone pancreatitis is usually due to an obstructing stone in the pancreatic duct near the sphincter of Oddi ( Bhatia M et al .,2005). In alcohol-related pancreatitis, it is believed that the acinar cells of the pancreas are susceptible to damage by ethanol and underlie the etiology of the disease ( Tonsi AF et al ., 2009). Another common cause, iatrogenic pancreatitis, may occur after endoscopic retrograde cholangiopancreatography (ERCP) in up to 5% of patients. Other etiologies of acute pancreatitis include medications, infections, trauma, hereditary, hypertriglyceridemia and autoimmune disease.

According to the American College of Gastroenterology, a patient must have two of the following three features present to make a diagnosis of acute pancreatitis The diagnostic criteria used for acute pancreatitis includes:

1. Clinical criteria - history of pain in abdomen radiating to the back and relieved on bending forward associated with tenderness/guarding in the upper abdomen.
2. Radiographic evidence - Computed Tomography findings suggestive of acute pancreatitis such as pancreatic edema, pancreatic necrosis, peripancreatic fluid collections
3. Biochemical - Serum amylase concentration greater than 180 Somogyii units (by the Somogyii method).

ELIGIBILITY:
Inclusion Criteria:

* 100 patients with acute pancreatitis admitted at Assiut university hospital and the diagnosis of acute pancreatitis is confirmed if at least two of the following three features present:

  1. abdominal pain characteristic of acute pancreatitis.
  2. serum amylase and/or lipase greater than 3 times the upper limit of normal .
  3. radiographically demonstrated acute pancreatitis on CT scan or abdominal ultrasound.

Exclusion Criteria:

1. Patients are excluded from the study if they do not meet the criteria for acute pancreatitis
2. Patients who are under the age of 16.
3. Patients with chronic pancreatitis.
4. Patients with recurrent acute pancreatitis

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Evaluation of the best prognostic parameter in patients with acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of the prognostic value of neutrophil _lymphocyte ratio in cbc in patients with acute pancreatitis admitted at assiut university hospitals. | one year
  evaluation of the prognostic value neutrophil lymphocyte ratio in patient with acute pancreatitis
evaluation of the prognostic value of LDH in patients with acute pancreatitis admitted at assiut university hospitals. | one year
  evaluation of the prognostic value of LDH ratio in patient with acute pancreatitis
evaluation of the prognostic value of urine analysis in patients with acute pancreatitis admitted at assiut university hospitals. | one year
  evaluation of the prognostic value of urine analysis ratio in patient with acute pancreatitis